CLINICAL TRIAL: NCT01252823
Title: Identification and Prevention of Sudden Cardiac Death Causes in Hemodialysis Patients
Brief Title: Implantable Loop Recorder in Hemodialysis Patients
Acronym: RYTHMODIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2010/33
Record Dates: First submitted 2010-11-04; First posted 2010-12-03 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Hemodialysis; Cardiac Arrhythmia; Cardiac Death
Keywords: Hemodialysis; Cardiac Arrhythmia; Cardiac Death; Implantable Loop Recorder
MeSH Terms: conditions — Arrhythmias, Cardiac; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implantable loop recorder (ILR) in hemodialysis patients (Experimental): implantation of loop recorder in hemodialysis patients
  Interventions: Device: Implantation of ILR

INTERVENTIONS:
Device: Implantation of ILR — Subcutaneous implantation of ILR under local anesthesia

SUMMARY:
The purpose of this study is to use implantable loop recorder (ILR) in patients under chronic hemodialysis to record arrhythmias and conduction disorders and correlate them with hemodialysis parameters.

DETAILED DESCRIPTION:
Primary cause of death in patients under chronic hemodialysis is Sudden Cardiac Death (SCD) (25% of all cause mortality). SCD is mainly due to cardiac arrhythmias (conduction disturbances or ventricular arrhythmias). These cardiac arrhythmias are highly sensitive to hydro-electrolytic disorders which are extremely frequent in patients under hemodialysis. In addition, other conditions leading to cardiac arrhythmias are frequent in this population such as ischemic myocardiopathy or dilated myocardiopathy. However, so far, little is known about the occurrence of arrhythmias because of studies using only standard Holter monitoring (24 to 48 hours monitoring at best).

The investigators sought to evaluate the incidence of cardiac arrhythmias by using an implantable loop recorder (ILR)(Reveal XT, Medtronic) that allows continuous rhythm monitoring for 24 months. This ILR will be implanted under local anesthesia.

Clinical follow-up will be performed during hemodialysis and rhythm management will be performed automatically using a remote-monitoring system (Carelink, Medtronic). Pre-programmed alerts (conduction disturbances, supra-ventricular arrhythmias or ventricular arrhythmias) recorded by the ILR will be sent automatically on a daily basis in our center. These data will be analyzed during week days from 9AM to 5PM. They will be reviewed by an electrophysiologists and depending on the potential lethality, the patients will be called and ask to come to the emergency room in case of high risk or the nephrologist will be contacted and he will see the patients during the next hemodialysis in case of on vital event.

ELIGIBILITY:
Inclusion Criteria:

* Patients under chronic hemodialysis
* Age between 45 and 80 yo
* written informed consent
* affiliated to the French Social Security system

Exclusion Criteria:

* Pace-maker or Implantable Cardioverter Defibrillator
* Active infection
* Neoplasia or any pathology with a life expectancy <12 months
* Cachexia
* Patient with restricted civic rights by law

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-12-28 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Occurrence of arrhythmia | Checked every days except Sundays and bank holidays during 24 Month
  * Type 1: Conduction disorders: 1A-Cardiac arrest, 1B-High degree AV Block, 1C-Sinus dysfunction (Sinus pause>3seconds, Bradycardia <30 bpm)
  * Type 2: Ventricular rhythm disorders ≥ 150 bpm: 2A-Polymorphic ventricular tachycardia, Torsades de pointe, Ventricular Fibrillation, 2B-Sustained ventricular tachycardia (>30 seconds), 2C- Non sustained ventricular tachycardia (>4 beats but <30 seconds)

SECONDARY OUTCOMES:
Study correlation between arrhythmic events (primary outcome) and hemodialysis parameters (general: day of dialysis, length of dialysis;clinical: weight variation during dialysis...; biological: potassium level, potassium variation...; ECG) | three times per weeks, at each hemodialysis
Incidence of supra-ventricular arrhythmia: 3A-Atrial Fibrillation, 3B-Atrial Tachycardia, 3C-Junctional tachycardia | Checked every days except Sundays and bank holidays during 24 Month

CONTACTS AND LOCATIONS:
Overall Officials: Christian COMBE, MD-PhD, Study Chair — University Hospital of Bordeaux, France; Antoine BENARD, MD, Study Chair — USMR, University Hospital of Bordeaux, France
Locations (9):
- France (9):
  - Clinique Saint Augustin, Bordeaux
  - University Hospital of Bordeaux, Bordeaux
  - Polyclinique Bordeaux-Nord Aquitaine, Bordeaux
  - CH de Haguenau, Haguenau
  - CH de Libourne, Libourne
  - CHU de Nantes, Nantes
  - CHU de Rennes, Rennes
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Derived] Sacher F, Jesel L, Borni-Duval C, De Precigout V, Lavainne F, Bourdenx JP, Haddj-Elmrabet A, Seigneuric B, Keller A, Ott J, Savel H, Delmas Y, Bazin-Kara D, Klotz N, Ploux S, Buffler S, Ritter P, Rondeau V, Bordachar P, Martin C, Deplagne A, Reuter S, Haissaguerre M, Gourraud JB, Vigneau C, Mabo P, Maury P, Hannedouche T, Benard A, Combe C. Cardiac Rhythm Disturbances in Hemodialysis Patients: Early Detection Using an Implantable Loop Recorder and Correlation With Biological and Dialysis Parameters. JACC Clin Electrophysiol. 2018 Mar;4(3):397-408. doi: 10.1016/j.jacep.2017.08.002. Epub 2017 Sep 27. PMID 30089568